CLINICAL TRIAL: NCT03867812
Title: Effect of Consumption of Different Foods on the Pharmacokinetics of a Small Dose of Ethanol: A Randomized Controlled, Clinical Trial in Healthy Individuals
Brief Title: Effect of Different Foods Together With a Small Dose of Alcohol on Alcohol Levels in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeno Functional Foods, LLC (Industry)
Collaborators: INQUIS Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: GIL-1842
Record Dates: First submitted 2019-03-05; First posted 2019-03-08 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Alcohol Use, Unspecified
MeSH Terms: conditions — Alcohol Drinking | interventions — Hazard Analysis and Critical Control Points

STUDY DESIGN:
Intervention Model Description: Open label, randomized, crossover, controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Fasting + alcoholic drink (No Intervention): No food (0 calories) but 250ml of water followed by an alcoholic drink (a 20% alcohol by volume cocktail dosed so that men receive 0.35g alcohol per kg of body weight and women a 0.30g/kg dose).
- SOBAR bar + alcoholic drink (Experimental): One 70g bar (210 calories) plus 250ml of water followed by an alcoholic drink (a 20% alcohol by volume cocktail dosed so that men receive 0.35g alcohol per kg of body weight and women a 0.30g/kg dose).
  Interventions: Other: SOBAR
- Control food + alcoholic drink (Active Comparator): 48.5g of General Mills Chexmix (Honey Nut Flavor, 210 calories) plus 250ml of water followed by an alcoholic drink (a 20% alcohol by volume cocktail dosed so that men receive 0.35g alcohol per kg of body weight and women a 0.30g/kg dose).
  Interventions: Other: Control food
- Full meal + alcoholic drink (Active Comparator): Stouffer's Bistro Crostini 5 Cheeses, Oikos Strawberry yogurt, Tropicana Orange juice, Dad's oatmeal cookie (635 calories total) followed by an alcoholic drink (a 20% alcohol by volume cocktail dosed so that men receive 0.35g alcohol per kg of body weight and women a 0.30g/kg dose).
  Interventions: Other: Full meal

INTERVENTIONS:
Other: SOBAR — SOBAR is a high protein nutrition bar optimized to delay gastric emptying
  Arms: SOBAR bar + alcoholic drink
Other: Control food — Chexmix (General Mills Inc.), Honey Nut Flavor
  Arms: Control food + alcoholic drink
Other: Full meal — Stouffer's Bistro Crostini 5 cheeses, Oikos Strawberry yogurt, Tropicana Orange juice, Dad's oatmeal cookie
  Arms: Full meal + alcoholic drink

SUMMARY:
Alcohol consumption is prevalent and frequently excessive and its use poses a major risk to both personal and public health. In the U.S., every month over 25% of adults and 40% of college students drink until their blood alcohol concentration (BAC) exceeds the legal limit of 0.08% and there is a great unmet need for interventions to help individuals better manage their BACs. Zeno Functional Foods has developed a protein bar, SOBAR, with the aim to control alcohol absorption when eaten prior to drinking. It is hypothesized that the SOBAR will slow stomach emptying resulting in a comparatively diminished peak BAC as well as a more stable BAC-time profile that is both safer and more pleasurable for the drinker.

DETAILED DESCRIPTION:
Alcohol consumption is not a new phenomenon; it has been part of human culture since the start of recorded time. As a consequence, advice on alcohol consumption is also not new with probably the best-known one by the Greek playwright Eubulus:

"Three bowls do I mix for the temperate: one to health, which they empty first; the second to love and pleasure; the third to sleep. When this bowl is drunk up, wise guests go home. The fourth bowl is ours no longer, but belongs to violence; the fifth to uproar; the sixth to drunken revel; the seventh to black eyes; the eighth is the policeman's; the ninth belongs to biliousness, and the tenth to madness and the hurling of furniture".

Moderate alcohol consumption appears to provide some protection against certain illnesses, including heart disease and diabetes, however counterbalancing this is that, simultaneously, alcohol consumption will also increase the risk of other serious diseases (Bagnardi et al, 2004; Di Castelnouvo et al, 2006; Djousse and Gaziano, 2008; Rehm et al, 2006; Standridge et al, 2004) as well as injury (Taylor et al, 2010). As the amount of alcohol usually consumed in a day increases, so does the risk of a wide range of physical and mental illnesses, including a number of cancers, liver disease and depression (Rehm et al, 2006).

As a consequence, the current advice as given by the USDA is not to consume alcohol at all and, when alcohol is consumed, it is to be done in moderation within a healthy eating pattern. These recommendations are consistent with the most recent review of global alcohol usage and the risks it poses (GBD 2016 Alcohol Collaborators, 2018).

Despite these guidelines, alcohol consumption is prevalent and frequently excessive and its use poses a major risk to both personal and public health. In the U.S., every month over 25% of adults and 40% of college students drink until their blood alcohol concentration (BAC) exceeds the legal limit of 0.08% and there is a great unmet need for interventions to help individuals better manage their BACs (www.niaaa.nih.gov/alcohol-health).

A person's maximal BAC, under a particular drinking scenario, is a result of many factors including how much alcohol they consumed, how quickly they consumed it, and the amount and characteristics of the food in their stomach. The contents of the stomach play a critical role in determining the alcohol absorption rate, and the maximal BAC, through their effect on the rate of gastric emptying (Holt, 1981). Furthermore, slower gastric emptying has been shown to increase the first pass metabolism of alcohol, both in the stomach as well as the liver, and can further diminish peak BAC (Oneta et al, 1998). Therefore, a food which has the ability to significantly slow the gastric emptying rate would be expected to significantly delay alcohol absorption, and due to increased first pass inactivation, limit the peak BAC as compared to drinking on an empty stomach. SOBAR is a high protein nutrition bar optimized to delay gastric emptying which has shown significant efficacy and safety in pilot studies.

Zeno Functional Foods ("ZENO") is an emerging company formed in January 2017 and headquartered in Redwood City, CA. ZENO's focus is on the development of functional foods for the improvement of public health. Their first product is a protein bar, SOBAR, developed with the aim to control alcohol absorption when eaten prior to drinking. It is hypothesized that the SOBAR will slow stomach emptying resulting in a comparatively diminished peak BAC as well as a more stable BAC-time profile that is both safer and more pleasurable for the drinker. In preliminary case studies, test subjects were given a defined cocktail after consuming either no food, a SOBAR prototype, a similarly caloric control food or a full meal, and the value of alcohol in the blood (BAC) was calculated from breath samples by a calibrated breathalyzer. BAC was lower after the SOBAR compared to having no food or comparable foods and were similar when compared to BAC levels after a full meal.

As the preliminary results were encouraging, a full clinical study using a similar paradigm to the case studies is now planned to explore the effect of SOBAR on BAC levels. The study will utilize an open-label, randomized controlled design and assess BAC indirectly from breath measurements using a calibrated breathalyzer. A calibrated breathalyzer is the standard method for an indirect measure of blood alcohol concentration and is well established to provide a reliable estimate of BAC, therefore, blood samples will not be collected.

PRIMARY OBJECTIVE:

To compare the maximal BAC concentration (BAC Cmax) estimated using a breathalyzer over 90 minutes after ingestion of a 20% by volume alcoholic drink after ingestion of either a SOBAR, an isocaloric control food, a full meal, or no food.

SECONDARY OBJECTIVES:

To compare the alcohol pharmacokinetics over 90 minutes (as measured by the IAUC60 and 90min) after ingestion of either a SOBAR, an isocaloric control food, a full meal, or when no food is consumed.

To compare the time to reach the maximal (BAC Tmax) using a breathalyzer after ingestion of either a SOBAR, an isocaloric control food, a full meal, or when no food is consumed.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating females, 25-65 years of age, inclusive
* Body mass index 20 - 30 kg/m2 inclusive
* Blood pressure: systolic < 140 and diastolic <95 mmHg.
* Social drinkers; average 2 or fewer drinks per day and have not had an episode of "binge drinking" over the previous 30 days. Binge drinking is defined has having 4 or more drinks (for women) / 5 or more drinks (for men) over the course of 2 hours. One drink is defined as either 5oz wine, 341ml of beer/cider or 1.5 oz. of distilled 80-proof spirit.
* Willing to maintain habitual diet, physical activity pattern, and body weight throughout the trial and consume the standard meal provided by GI Labs the evening before each test day
* Subject is willing to abstain from strenuous exercise, alcoholic drinks, and cannabis use 24hours before study visits.
* Subject is willing to refrain from driving or operating any vehicle when leaving GI Labs after the test visit
* Subject is willing to sign on each test day a statement acknowledging that the subject is aware that he/she has consumed alcohol that morning
* Willing to maintain current dietary supplement use throughout the trial. On test days, subject agrees not to take any dietary supplements or caffeine. Failure to comply will result in a rescheduled test visit.
* No major illness or surgery requiring hospitalization within 3 months of the first study visit after screening.
* No history of cardiovascular, metabolic, respiratory, renal, gastrointestinal or hepatic disease.
* Subjects must be eligible to receive income in Canada and be covered by a health insurance such as OHIP.
* Absence of health conditions that would prevent fulfillment of study requirements as judged by the Investigator on the basis of medical history.
* Understanding the study procedures and willing to provide informed consent to participate in the study and authorization to release relevant protected health information to the study investigator.
* Female subjects are willing to use a contraceptive method to avoid pregnancy during the study period. Willing to take a urine pregnancy test the day of each study.

Exclusion Criteria:

* Failure to meet all the inclusion criteria
* Smoker
* Known history of gastrointestinal, liver, kidney, or cardiovascular (including but not limited to atherosclerotic disease, history of myocardial infarction, peripheral arterial disease, stroke), and pulmonary disease
* History of mental disease, seizures, use or abuse of psychoactive medications (including but not limited to cocaine, amphetamines, opiates, sedatives, benzodiazepines, and hallucinogens) or any medication or condition which might, in the opinion of Dr. Wolever, the medical director of GI labs, either: 1) make participation dangerous to the subject or to others, or 2) affect the results.
* Use of antibiotics within 4 weeks of start of study.
* History or diagnosis of alcohol use disorder or binge drinking (4 or more drinks for women and 5 or more drinks for men within a 2-hour window) as defined by the current NIAAA guidelines.
* Major trauma or surgical event within 3 months of screening.
* Of East Asian descent or having a history of alcohol induced flushing reaction.
* Unwillingness or inability to comply with the experimental procedures and to follow GI Labs safety guidelines.
* Known intolerance, sensitivity or allergy to any ingredients in the study products.
* Extreme dietary habits as judged by the Investigator (i.e. Atkins diet, very high protein diets, etc).
* Change in body weight of >3.5kg within 4 weeks of the screening visit.
* Presence of any signs or symptoms of an active infection within 5 d prior to any test visit. If an infection occurs during the study period, test visits should be rescheduled until all signs and symptoms have resolved and any treatment (i.e. antibiotic therapy) has been completed at least 5 d prior to each test visit.
* History of cancer in the prior two years, except for non-melanoma skin cancer.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Maximal blood alcohol concentration (BAC Cmax) | 90 minutes
  As measured indirectly using a breathalyzer, the level of peak BAC during the experimental timeframe.

SECONDARY OUTCOMES:
Incremental area under the curve at 60min (IAUC 60) | 60 minutes
  As measured indirectly using a breathalyzer, the incremental area under the BAC vs time curve over the experimental timeframe.
Incremental area under the curve at 90min (IAUC 90) | 90 minutes
  As measured indirectly using a breathalyzer, the incremental area under the BAC vs time curve over the experimental timeframe.
Time to reach maximal blood alcohol concentration (BAC Tmax) | 90 minutes
  As measured indirectly using a breathalyzer, the time from the start of consuming the alcohol until the peak BAC is reached during the experimental timeframe.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Wolever, D.M., Ph.D., Principal Investigator — INQUIS Clinical Research
Locations (1):
- INQUIS Clinical Research Ltd., Toronto, Ontario, Canada

REFERENCES:
- [Background] Di Castelnuovo A, Costanzo S, Bagnardi V, Donati MB, Iacoviello L, de Gaetano G. Alcohol dosing and total mortality in men and women: an updated meta-analysis of 34 prospective studies. Arch Intern Med. 2006 Dec 11-25;166(22):2437-45. doi: 10.1001/archinte.166.22.2437. PMID 17159008
- [Background] Djousse L, Gaziano JM. Alcohol consumption and heart failure: a systematic review. Curr Atheroscler Rep. 2008 Apr;10(2):117-20. doi: 10.1007/s11883-008-0017-z. PMID 18417065
- [Background] Bagnardi V, Zambon A, Quatto P, Corrao G. Flexible meta-regression functions for modeling aggregate dose-response data, with an application to alcohol and mortality. Am J Epidemiol. 2004 Jun 1;159(11):1077-86. doi: 10.1093/aje/kwh142. PMID 15155292
- [Background] Rehm, J., Ballunas, D., Broschu, S., Fischer, B., Gnam, W. & Patras, J., et al. (2006a). The Costs of Substance Abuse in Canada, 2002. ISBN: 1-897321-10-4 (CD-ROM). Ottawa: Canadian Centre on Substance Abuse.
- [Background] Standridge JB, Zylstra RG, Adams SM. Alcohol consumption: an overview of benefits and risks. South Med J. 2004 Jul;97(7):664-72. doi: 10.1097/00007611-200407000-00012. PMID 15301124
- [Background] Taylor B, Irving HM, Kanteres F, Room R, Borges G, Cherpitel C, Greenfield T, Rehm J. The more you drink, the harder you fall: a systematic review and meta-analysis of how acute alcohol consumption and injury or collision risk increase together. Drug Alcohol Depend. 2010 Jul 1;110(1-2):108-16. doi: 10.1016/j.drugalcdep.2010.02.011. Epub 2010 Mar 16. PMID 20236774
- [Background] GBD 2016 Alcohol and Drug Use Collaborators. The global burden of disease attributable to alcohol and drug use in 195 countries and territories, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet Psychiatry. 2018 Dec;5(12):987-1012. doi: 10.1016/S2215-0366(18)30337-7. Epub 2018 Nov 1. PMID 30392731
- [Background] Holt S. Observations on the relation between alcohol absorption and the rate of gastric emptying. Can Med Assoc J. 1981 Feb 1;124(3):267-77, 297. PMID 7459787
- [Background] Oneta CM, Simanowski UA, Martinez M, Allali-Hassani A, Pares X, Homann N, Conradt C, Waldherr R, Fiehn W, Coutelle C, Seitz HK. First pass metabolism of ethanol is strikingly influenced by the speed of gastric emptying. Gut. 1998 Nov;43(5):612-9. doi: 10.1136/gut.43.5.612. PMID 9824340